CLINICAL TRIAL: NCT01250405
Title: Acute Effects of Cinacalcet on Arterial Stiffness and Ventricular Function in Hemodialysis Patients
Acronym: ECIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Karine Marquis, Professionnelle de recherche, Laval University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CA2009-0008
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinacalcet (Active Comparator)
  Interventions: Drug: Cinacalcet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — One sequence receives Cinacalcet 30mg /d for 7 days followed by placebo for 7 days
  Arms: Cinacalcet
Drug: Placebo — One sequence receives placebo for 7 days followed by Cinacalcet 30mg/d for 7 days
  Arms: Placebo

SUMMARY:
The primary objective is to determine whether reduction of serum calcium concentration by cinacalcet leads to reduction of mean blood pressure adjusted c-fPWV. The secondary objectives are to study the effects of calcium reduction on 1) carotid-radial PWV (c-rPWV), 2) common carotid artery (CCA) biomechanics, 3) pulse wave profile and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* chronic (> 3 months) hemodialysis population of > 18 years old
* PTH > 300 ng/L
* corrected Ca > 2.10 mmol/L
* stable hypertensive drugs (> 1 month)
* stable doses of phosphate binders and dialysis calcium concentration
* palpable femoral pulse
* systolic BP of 90-180 mmHg
* expected survival of > 6 months

Exclusion Criteria:

* hemodialysis > 3 years
* acute infection
* history of myocardial infarction or stroke within the past 3 months
* inability to consent
* intolerance to cinacalcet
* inadequate birth control

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | Arterial stiffness with be measured after 1 week with placebo and after 1 week with cinacalcet

SECONDARY OUTCOMES:
Ventricular function | Ventricular function with be measured after 1 week with placebo and after 1 week with cinacalcet

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Agharazii, MD, Principal Investigator — Laval University
Locations (1):
- Karine Marquis, Québec, Quebec, Canada

REFERENCES:
- [Derived] Poulin A, Bellemare PL, Fortier C, Mac-Way F, Desmeules S, Marquis K, Gaudreault V, Lebel M, Agharazii M. Acute effects of cinacalcet on arterial stiffness and ventricular function in hemodialysis patients: A randomized double-blinded crossover study. Medicine (Baltimore). 2017 May;96(21):e6912. doi: 10.1097/MD.0000000000006912. PMID 28538380